CLINICAL TRIAL: NCT02038725
Title: MIDNOR-TIA - a Prospective Cohort Study of 600 TIA Patients in Central Norway
Brief Title: MIDNOR-TIA - a Study of 600 Patients With Transient Ischemic Attack
Acronym: MIDNOR-TIA
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1224
Record Dates: First submitted 2013-12-28; First posted 2014-01-16 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2019-05

CONDITIONS: Ischemic Attack, Transient; Stroke
Keywords: Risks; Risk Factors; ABCD2 score; Predictive Value of Tests; Risk Assessment; Severity of Illness Index; Decision Support Techniques
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIA in last 2 weeks

SUMMARY:
Patients with a transient ischemic attack (TIA) are at high risk of stroke. Rapid assessment and treatment can reduce the risk. Several international guidelines recommend a test, the ABCD2 score, to identify TIA patients with low and high risk for stroke. The main purpose of this study is to investigate stroke risk after TIA in both short (1 week) and long term (3 months/1 year), and to assess whether the ABCD2 score ('Age, blood pressure, clinical features, duration of TIA, diabetes score) is an adequate tool for predicting stroke risk. Secondary aims are to explore whether adopting imaging modalities (ultrasound, MRI) and biological markers of blood into a risk score could improve the predictive value of the ABCD2 score and still be feasible in a daily clinical practice. Further on overall risk factors in TIA patients, and the incidence of other vascular events will be studied. A substudy designed as a randomised controlled trial evaluates pharmaceutical counseling in a subset of participants. Cost-benefit analysis, and a long-term follow-up (5 years) is planned.

ELIGIBILITY:
Inclusion Criteria:

* Probable or possible transient ischemic attack
* Residing in Central Norway
* Examined within 2 weeks after the onset of symptoms
* Modified Rankin Scale 3 or less and living at home
* Informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a hospital in Central Norway with a recent probable or possible transient ischemic attack
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting with stroke within 1 week after transient ischemic attack | 1 week
  Measured by using data from the Norwegian Stroke Registry

SECONDARY OUTCOMES:
Number of patients presenting with stroke within 3 months after transient ischemic attack | 3 months
  Measured by using data from the Norwegian Stroke Registry
Correlation between the ABCD2 score and the incidence of stroke within 1 week after transient ischemic attack | 1 week
  Measured by comparing the ABCD2 score and the incidence of stroke within 1 week after transient ischemic attack based on data from the Norwegian Stroke Registry
Correlation between the ABCD2 score and the incidence of stroke within 3 months after transient ischemic attack | 3 months
  Measured by comparing the ABCD2 score and the incidence of stroke within 3 months after transient ischemic attack based on data from the Norwegian Stroke Registry
Incidence of other vascular events within 1 week after transient ischemic attack | 1 week
  Measured by using data from national health registries
Cost-benefit analysis | 1 year
  Economic analysis that compares the costs of admission to hospital versus outpatient assessment of patients who have had transient ischemic attacks
Number of patients presenting with stroke within 1 year after transient ischemic attack | 1 year
  Measured by using data from the Norwegian Stroke Registry
Correlation between the ABCD2 score and the incidence of stroke within 1 year after transient ischemic attack | 1 year
  Measured by comparing the ABCD2 score and the incidence of stroke within 1 year after transient ischemic attack based on data from the Norwegian Stroke Registry
Incidence of other vascular events within 3 months after transient ischemic attack | 3 months
  Measured by using data from national health registries
Incidence of other vascular events within 1 year after transient ischemic attack | 1 year
  Measured by using data from national health registries

CONTACTS AND LOCATIONS:
Overall Officials: Bent Indredavik, PhD, Prof, Study Director — Norwegian University of Science and Technology
Locations (8):
- Norway (8):
  - Ålesund Sykehus, Ålesund
  - Kristiansund Sykehus, Kristiansund
  - Levanger Sykehus, Levanger
  - Molde Sykehus, Molde
  - Namsos Sykehus, Namsos
  - Orkdal Sykehus, Orkanger
  - St Olavs Hospital, Trondheim
  - Volda Sykehus, Volda

REFERENCES:
- [Result] Ildstad F, Ellekjaer H, Fjaertoft H, Indredavik B. MIDNOR TIA - a prospective cohort study of 586 patients, baseline data from a subgroup of 363 patients examined with diffusion-weighted imaging. International Journal of Stroke 10(suppl 2):242, 2015 (Meeting Abstract ESOC-1527)
- [Result] Ildstad F, Ellekjaer H, Wethal T, Lydersen S, Sund JK, Fjaertoft H, Schuler S, Horn JW, Brathen G, Midtsaether AG, Morsund AH, Lillebo ML, Seljeseth YM, Indredavik B. Stroke risk after transient ischemic attack in a Norwegian prospective cohort. BMC Neurol. 2019 Jan 3;19(1):2. doi: 10.1186/s12883-018-1225-y. PMID 30606138
- [Result] Ildstad F, Ellekjaer H, Wethal T, Lydersen S, Fjaertoft H, Indredavik B. ABCD3-I and ABCD2 Scores in a TIA Population with Low Stroke Risk. Stroke Res Treat. 2021 Feb 25;2021:8845898. doi: 10.1155/2021/8845898. eCollection 2021. PMID 33708373